CLINICAL TRIAL: NCT02841267
Title: A Phase 1b/2, Open-Label, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of PF-06252616 in Ambulatory Participants With LGMD2I
Brief Title: A Trial of PF-06252616 in Ambulatory Participants With LGMD2I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kathryn Wagner (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Kathryn Wagner, Director, Center for Genetic Muscle Disorders, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Organization: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WI203720
Record Dates: First submitted 2016-07-12; First posted 2016-07-22 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: LGMD2I
MeSH Terms: conditions — Muscular Dystrophy, Limb-Girdle, Type 2I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose, Cohort 1 (Active Comparator): 4 subjects will be enrolled in cohort 1 and will receive an initial dose of 5mg/kg PF 06252616 IV every 4 weeks. Following 32 weeks of treatment and a safety review, if no stopping rules have been met, subjects will be receive an additional 32 weeks of treatment with 40 mg/kg PF 06252616 IV every 4 weeks.
  Interventions: Drug: PF 06252616
- Middle dose, Cohort 2 (Active Comparator): 8 subjects will be enrolled in cohort 2 and receive 20 mg/kg of PF 06252616 IV every 4 weeks for 32 weeks.
  Interventions: Drug: PF 06252616
- High dose, Cohort 3 (Active Comparator): 8 subjects will be enrolled in cohort 3 and receive 40 mg/kg of PF06252616 IV every 4 weeks for 32 weeks.
  Interventions: Drug: PF 06252616

INTERVENTIONS:
Drug: PF 06252616

SUMMARY:
The investigational product PF 06252616, a humanized anti myostatin monoclonal antibody that neutralizes myostatin (GDF8) is in development for the treatment of Limb Girdle Muscular Dystrophy 2I (LGMD2I) to preserve and/or improve muscle function.

This study will provide the clinical assessment of the safety, tolerability, Pharmacokinetics and Pharmacodynamics of PF 06252616 following repeat IV doses in ambulatory adults with LGMD2I.

DETAILED DESCRIPTION:
This study is a Phase 1b/2, open-label multiple ascending dose escalation study to evaluate the safety, tolerability, efficacy, PK and PD of PF 06252616 in ambulatory adults with LGMD2I. The study design is intended to determine the optimal safe and pharmacologically active dose of PF 06252616 in LGMD2I while providing an opportunity for all subjects to receive active drug for a rare and disabling disorder. The study will be conducted in three periods: Lead-In, Treatment and Follow-up periods. The Lead-In and Follow-up periods will each be 16 weeks to allow an assessment of the change of various outcome measures of this period of time and comparison of change in function before, during and after treatment. The Treatment period will be 32 weeks. Three cohorts of participants will be enrolled and receive escalating doses of PF 06252616. The first cohort will have the option to crossover to the highest dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age ≥ 18
2. Diagnosis of LGMD2I as defined by clinical presentation consistent with LGMD2I and FKRP gene testing showing biallelic alterations known or likely to be pathogenic. Diagnosis must be confirmed in subject's medical history and by genetic testing obtained during routine clinical care for diagnostic purposes as reported from an appropriate regulated laboratory using a clinically validated genetic test (genetic testing is not provided by the sponsor).
3. Ability to walk/run 10m
4. Ability to rise from chair
5. Adequate hepatic and renal function on screening laboratory assessments
6. Iron content estimate on the screening liver MRI within the normal range as determined by R2* value (R2* ≤ 139 Hz at 3.0T).
7. Participant must provide written informed consent for participating in study.
8. Participant must possess the ability, per the Principal Investigator (PI), to understand and comply with protocol instruction for the entire duration of the study.

Exclusion Criteria:

1. Known cognitive impairment or behavioral issues that would impede the ability to provide informed consent or to follow study instructions.
2. History of major surgical procedure within 6 weeks of signing the informed consent or planned surgery during the study.
3. Any injury which may impact functional testing. Previous injuries must be fully healed prior to consent. Prior lower limb fractures must be fully healed and at least 3 months from injury dates.
4. Previous treatment with another investigational product within 30 days or 5 half-lives, (whichever is longer) prior to consenting.
5. Corticosteroid treatment within 3 months prior to consenting.
6. Compromised cardiac function (left ventricular ejection fraction <50%).
7. Unwilling or unable (e.g. metal implants, requires sedation) to undergo examination with closed MRI without sedation.
8. History of allergic or anaphylactic reaction to a therapeutic or diagnostic protein.
9. Female subjects who are pregnant or nursing.
10. Subjects who, are biologically capable of having children who are unwilling or unable to use highly effective methods of contraception (as outlined in this protocol) during sexual activity for the duration of the study and through completion of final study visit.
11. Predisposition to iron accumulation. (Serum iron >1.2 X ULN, serum ferritin >1.2 ULNN).
12. Underlying disposition for bleeding disorder on screening laboratory assessment (PT/INR>1.25 X ULN, aPTT > 1.25 ULN, fecal occult blood is positive)
13. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic, or allergic disease.
14. Unwillingness or inability to comply with the requirements of this protocol (in the opinion of the PI) including, but not limited to, the presence of any condition (physical, mental, or social) that is likely to affect the participant's ability to return for study visits or adhere to the visit schedule.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-07; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn R Wagner, MD/PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Hugo W. Moser Research Institute at Kennedy Krieger, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung DG, Bocchieri AE, Ahlawat S, Jacobs MA, Parekh VS, Braverman V, Summerton K, Mansour J, Bibat G, Morris C, Marraffino S, Wagner KR. Longitudinal functional and imaging outcome measures in FKRP limb-girdle muscular dystrophy. BMC Neurol. 2020 May 19;20(1):196. doi: 10.1186/s12883-020-01774-5. PMID 32429923

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant in Cohort 2 was consented, but elected to withdraw from the study prior to assignment to a treatment arm.
Groups:
- Low Dose, Cohort 1: 4 subjects will be enrolled in cohort 1 and will receive an initial dose of 5mg/kg PF 06252616 IV every 4 weeks. Following 32 weeks of treatment and a safety review, if no stopping rules have been met, subjects will be receive an additional 32 weeks of treatment with 40 mg/kg PF 06252616 IV every 4 weeks.
  PF 06252616
- Middle Dose, Cohort 2: 8 subjects will be enrolled in cohort 2 and receive 20 mg/kg of PF 06252616 IV every 4 weeks for 32 weeks.
  PF 06252616
- High Dose, Cohort 3: 8 subjects will be enrolled in cohort 3 and receive 40 mg/kg of PF06252616 IV every 4 weeks for 32 weeks.
  PF 06252616
Period: Lead-in (Untreated)
Arm/Group | Low Dose, Cohort 1 | Middle Dose, Cohort 2 | High Dose, Cohort 3
Started (Participants were observed for 16 weeks prior to treatment.) | 4 | 7 | 8
Completed | 4 | 7 | 8
Not Completed | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Low Dose, Cohort 1 | Middle Dose, Cohort 2 | High Dose, Cohort 3
Started | 4 (Cohort 1 was invited to continue receiving 40mg/kg of study drug every 4 weeks for 28 weeks.) | 7 | 8
Completed | 4 | 7 | 8
Not Completed | 0 | 0 | 0
Period: Extension Study
Arm/Group | Low Dose, Cohort 1 | Middle Dose, Cohort 2 | High Dose, Cohort 3
Started | 4 (Cohort 1 was invited to continue receiving 40mg/kg of study drug every 4 weeks for 28 weeks.) | 6 (Cohort 2 was invited to continue receiving 40mg/kg of study drug every 4 weeks for 40 weeks.) | 6 (Cohort 3 was invited to continue receiving 40mg/kg of study drug every 4 weeks for 24 weeks.)
Completed | 4 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Target enrollment was reached for Cohort 1 and Cohort 3. For Cohort 2, 8 subjects were screened, but 1 voluntarily withdrew prior to enrollment and was not replaced.
Groups:
- Cohort 1 - Low Dose: 4 subjects were enrolled in cohort 1 and received an initial dose of 5mg/kg PF 06252616 IV every 4 weeks. Following 32 weeks of treatment, subjects received an additional 32 weeks of treatment with 40 mg/kg PF 06252616 IV every 4 weeks.
- Cohort 2 - Middle Dose: 7 subjects were enrolled in cohort 2 and received 20 mg/kg of PF 06252616 IV every 4 weeks for 32 weeks.
- Cohort 3 - High Dose: 8 subjects were enrolled in cohort 3 and received 40 mg/kg of PF06252616 IV every 4 weeks for 32 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose | Total
Number analyzed (Participants) | 4 | 7 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (8) | 41 (18) | 34 (9.9) | 39 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 12
  Male | 1 | 3 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 7 | 8 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting or Intolerability Treatment Related Adverse Events
Description: Adverse events include subject-reported symptoms as well as clinically-significant changes in laboratory testing, vital signs, and suicide screening (based on the Columbia Suicide Severity Rating Scale).
Time Frame: Baseline through 64 weeks
Population: All enrolled subjects are included in the analysis.
Measure: Number; unit: events
Groups:
- Cohort 1: 4 subjects received 32 weeks of treatment with 5mg/kg PF 06252616 IV every 4 weeks followed by an additional 32 weeks of treatment with 40 mg/kg PF 06252616 IV every 4 weeks.
- Cohort 2, Middle Dose: 7 subjects were enrolled in cohort 2 and received 20 mg/kg of PF 06252616 IV every 4 weeks for 32 weeks.
- Cohort 3, High Dose: 8 subjects were enrolled in cohort 3 and received 40 mg/kg of PF06252616 IV every 4 weeks for 32 weeks.
Arm/Group | Cohort 1 | Cohort 2, Middle Dose | Cohort 3, High Dose
Number analyzed (Participants) | 4 | 7 | 8
events
  Any adverse event | 45 | 21 | 40
  Serious adverse event | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Serum Concentration at Steady State (Cmax, ss) of GDF-8
Description: The concentration of myostatin (GDF-8) was measured in serum 2 hours after dose administration at two visits (Day 337 and Day 393 for Cohort 1; Day 113 and 169 for Cohorts 2 and 3)where drug concentration had reached steady state. The highest concentration from these two time points was averaged for each cohort.
Time Frame: Day 337 and Day 393 for Cohort 1; Day 113 and 169 for Cohorts 2 and 3
Population: All enrolled participants were analyzed. For Cohort 1, measurements are provided for the 40mg/kg dosing period.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Cohort 1 - Low Dose: 4 subjects were enrolled in cohort 1 and received an initial dose of 5mg/kg PF 06252616 IV every 4 weeks. Following 32 weeks of treatment and a safety review, subjects received an additional 32 weeks of treatment with 40 mg/kg PF 06252616 IV every 4 weeks.
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
ng/ml | 9.02 (3.20) | 8.96 (3.02) | 9.67 (6.45)

3. Secondary Outcome: Minimum Observed Serum Trough Concentration at Steady State (Ctrough,ss) of GDF-8
Description: The concentration of myostatin (GDF-8) was measured in serum prior to dose administration at two time points (Day 337 and Day 393 for Cohort 1; Day 113 and 169 for Cohorts 2 and 3) where drug concentration had reached steady state. The lowest concentration from these two time points was averaged for each cohort.
Time Frame: Day 337 and Day 393 for Cohort 1; Day 113 and 169 for Cohorts 2 and 3
Population: All enrolled participants were analyzed. For Cohort 1, measurements are provided for the 40mg/kg dosing period.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
ng/ml | 8.80 (2.96) | 9.68 (2.21) | 9.78 (7.61)

4. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-06252616
Description: The peak concentration of study drug (PF-06252616) was measured in serum following dose administration at two time points (Day 113 and Day 169) where drug concentration had reached steady state. The higher concentration from these two time points was averaged for each cohort.
Time Frame: Day 113 and Day 169
Population: All enrolled participants were analyzed. For Cohort 1, measurements are provided for 5mg/kg dosing period.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
ng/ml | 215306.5 (29490.4) | 779015.7 (115450.0) | 1625203 (271159.6)

5. Secondary Outcome: Minimum Observed Serum Trough Concentration (Ctrough) of PF-06252616
Description: The peak concentration of study drug (PF-06252616) was measured in serum prior to dose administration at two time points (Day 113 and Day 169) where drug concentration had reached steady state. The lower concentration from these two time points was averaged for each cohort.
Time Frame: Day 113 and Day 169
Population: All enrolled participants were analyzed. For Cohort 1, measurements are provided for the 5mg/kg dosing period.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 7
ng/ml | 67016.8 (25887.3) | 224024.1 (58734.5) | 408814.1 (96607.6)

6. Secondary Outcome: Immunogenicity: Incidence of Anti-drug Antibody
Description: Blood samples were tested for the presence of anti-drug antibodies prior to the initiation of study drug, at dose escalation (Cohort 1 only), and at 3 separate time points after the last dose was given.
Time Frame: Baseline through 96 weeks
Population: All enrolled subjects were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
Participants | 0 | 0 | 0

7. Secondary Outcome: Mean Change From Baseline in 10 Meter Walk/Run Time in Seconds
Description: Subjects are asked to run or walk as quickly as possible for 10 meters from a standing position. The total time to traverse 10 meters is recorded in seconds.
Time Frame: Baseline through 32 weeks
Population: All enrolled subject were included in the analysis. For Cohort 1, data is provided for the 5mg/kg dosing period.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
seconds | 1.60 (2.95) | -0.09 (0.11) | 0.18 (0.31)

8. Secondary Outcome: Mean Change From Baseline of Forced Vital Capacity in Liters
Description: The total forced vital capacity was measured using a bedside spirometer. The best of 3 trials was recorded.
Time Frame: Baseline through 32 weeks
Population: All enrolled subjects were included in the analysis. For Cohort 1, data is provided for the 5mg/kg dosing period.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
liters | 0.03 (0.14) | 0.02 (0.15) | -0.05 (0.14)

9. Secondary Outcome: Mean Change From Baseline in 2MWD in Meters
Description: Average change in distance (in meters) walked in 2 minutes.
Time Frame: Baseline through 32 weeks
Population: All enrolled participants were analyzed. For Cohort 1, measurements are provided for the 5mg/kg dosing period.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
meters | -4.25 (9.91) | 2.00 (7.77) | 2.13 (5.17)

10. Secondary Outcome: Mean Change From Baseline in TUG in Seconds
Description: The timed-up-and-go test (TUG) is the total time it takes the subject to rise from a seated position, walk to a marker 3 meters away, return to the chair, and sit.
Time Frame: Baseline through 32 weeks
Population: All enrolled subjects are included in the analysis. For Cohort 1, data is provided for the 5mg/kg dosing period.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
seconds | 0.67 (1.15) | 0.29 (1.11) | -0.50 (1.51)

11. Secondary Outcome: Mean Change From Baseline in Muscle Strength as Measured by Modified MRC Scale
Description: Twenty-two muscle groups were measured on a modified MRC scale ranging from 1 through 12. The total scores from all 22 muscle groups were added to generate a summary score ranging from 12 to 264 with higher scores signifying greater strength. The change in summary score was calculated over the first 32 weeks of treatment.
Time Frame: Baseline through 32 weeks
Population: All enrolled participants were analyzed after 32 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 4 | 7 | 8
score on a scale | 9.75 (6.18) | 7.57 (8.62) | 2.43 (4.54)

ADVERSE EVENTS:
Time Frame: Baseline through 124 weeks
Description: Subject reported adverse events, as well as clinically relevant changes in laboratory screening, physical examination, suicide screening, cardiac screening are reported.
Groups:
- Lead-in: All subjects were observed in a 16-week untreated lead-in-phase prior to allocation to dosing cohorts.
- Cohort 1 - Low Dose: Subjects received an initial dose of 5mg/kg PF 06252616 IV every 4 weeks for 32 weeks.
- Cohort 1 - High Dose: Following the Low Dose period, subjects in Cohort 1 received an additional 32 weeks of treatment with 40 mg/kg PF 06252616 IV every 4 weeks.
- Cohort 1 Extension: Subjects enrolled in Cohort 1 were given the option to receive PF 06252616 at 40 mg/kg every 4 weeks for an additional 28 weeks.
- Cohort 2: Subjects received 20 mg/kg of PF 06252616 IV every 4 weeks for 32 weeks.
- Cohort 2 Extension: Subjects enrolled in Cohort 2 were given the option to receive PF 06252616 at 40 mg/kg every 4 weeks for an additional 40 weeks.
- Cohort 3: Subjects received 40 mg/kg of PF 06252616 IV every 4 weeks for 32 weeks.
- Cohort 3 Extension: Subjects enrolled in Cohort 3 were given the option to receive PF 06252616 at 40 mg/kg every 4 weeks for an additional 24 weeks.
Arm/Group | Lead-in | Cohort 1 - Low Dose | Cohort 1 - High Dose | Cohort 1 Extension | Cohort 2 | Cohort 2 Extension | Cohort 3 | Cohort 3 Extension
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/4 | 0/4 | 0/4 | 0/7 | 0/6 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/4 | 0/4 | 0/4 | 0/7 | 1/6 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 9/19 | 4/4 | 4/4 | 4/4 | 6/7 | 4/6 | 7/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in (N=19) | Cohort 1 - Low Dose (N=4) | Cohort 1 - High Dose (N=4) | Cohort 1 Extension (N=4) | Cohort 2 (N=7) | Cohort 2 Extension (N=6) | Cohort 3 (N=8) | Cohort 3 Extension (N=6)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in (N=19) | Cohort 1 - Low Dose (N=4) | Cohort 1 - High Dose (N=4) | Cohort 1 Extension (N=4) | Cohort 2 (N=7) | Cohort 2 Extension (N=6) | Cohort 3 (N=8) | Cohort 3 Extension (N=6)
Pain associated with muscle biopsy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Numbness following biopsy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower extremity edema following biopsy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin avulsion following biopsy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intravenous catheter infiltration (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis at IV site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall - not otherwise specified (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain post fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Fracture - pelvic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee injury post fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder injury post fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial injury post fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle injury post fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shoulder pain - not otherwise specified (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee pain - not otherwise specified (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain - not otherwise specified (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip pain - not otherwise specified (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Worsening cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory symptoms (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 3 (3) | 0 (0) | 2 (5) | 1 (1)
Flu-like illness (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Environmental allergies (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious illness - not otherwise specified (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic hypertrophy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaginal yeast infection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision abnormality - not otherwise specified (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye twitching (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash - not otherwise specified (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sore (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst - not otherwise specified (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Greater than 5% of baseline weight
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Greater than 5% of baseline weight
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketones detected in urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cells in urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated serum iron levels (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Low serum iron levels (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Elevated amylase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated serum ferritin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low serum ferritin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoccult positive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
New diagnosis - carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
New diagnosis - hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
New diagnosis - umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
New diagnosis - bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
New diagnosis - personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02841267/ICF_000.pdf
  • Study Protocol (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT02841267/Prot_001.pdf
  • Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT02841267/SAP_002.pdf